CLINICAL TRIAL: NCT02077738
Title: High-frequency Chest Wall Oscillation in Prolonged Mechanical Ventilation Patients-a Randomized Controlled Trial
Brief Title: HFCWO in Prolonged Mechanical Ventilation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C10216; huang5598 (Other: Taichung VGH)
Record Dates: First submitted 2014-02-20; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Ventilator Dependency
Keywords: effectiveness; elderly; high frequency chest wall oscillation; mechanical ventilation; pneumonia; randomized controlled trial
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFCWO (Experimental): HFCWO for 15 min twice a day
  Interventions: Device: HFCWO (Hill-Rom Vest™ Airway Clearance System)
- placebo (Placebo Comparator): not to receive high-frequency chest wall oscillation (HFCWO)

INTERVENTIONS:
Device: HFCWO (Hill-Rom Vest™ Airway Clearance System) — study subjects in the HFCWO group received HFCWO for 15 min twice a day for 5 days after extubation
  Other Names: Hill-Rom Vest™ Airway Clearance System
  Arms: HFCWO

SUMMARY:
The effectiveness, safety and tolerance/comfort of high-frequency chest wall oscillation (HFCWO) in prolonged mechanical ventilation patients remain unknown. This study aimed to test the hypothesis that HFCWO could produce greater clearance volume of sputum, greater improvement rates in serial changes in the chest X-ray (CXR), and greater weaning success rates after extubation in Prolonged Mechanical Ventilation (PMV) patients with intra-tracheal intubation.

DETAILED DESCRIPTION:
For over 20 years, studies have attempted to examine the effectiveness, safety and tolerance/comfort of HFCWO in the management of surgical and non-surgical patients who had impaired bronchial secretion clearance, including those with neuromuscular disorders, chronic obstructive pulmonary disease, cystic fibrosis, and blunt thoracic trauma, or those hospitalized for critical cardiac/abdominal/thoracic surgery. However, these outcomes of HFCWO on PMV patients remain unknown.

This parallel-design, randomized controlled trial aimed to test the hypothesis that HFCWO could produce greater clearance volume of sputum, greater improvement rates in serial changes in the chest X-ray (CXR), and greater weaning success rates after extubation in PMV patients with intra-tracheal intubation. Moreover, the safety and tolerance/comfort of HFCWO in PMV patients after removal of endotracheal tubes were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. continuous intra-tracheal intubation and mechanical ventilator support for at least 21 days
2. age ≥20 year-old
3. having an acute or chronic pulmonary condition requiring secretion mobilization as judged by the physician
4. alert consciousness; completion of the Modified Borg Scale (MBS) and Hamilton Anxiety Scale (HAS)
5. scheduled extubation within 24 hours after enrollment
6. without any contraindication for HFCWO (i.e., recent spinal injuries which have not yet been stabilized and active hemorrhage with hemodynamic instability)

Exclusion Criteria:

1. those who had undergone tracheostomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness as determined by weaning success rates | up to 5 days after extubation
  Successful weaning was defined as continuous liberation from mechanical ventilator support longer than 5 days.
Effectiveness as determined by daily clearance volume of sputum | up to 5 days after extubation
  The daily clearance volume of sputum was determined by the numbers of sputum suction per day
Effectiveness as determined by serial changes in sputum coloration | up to 5 days after extubation
  The sputum coloration was determined by the Color Card for Body Fluid (CCBF). The CCBF was designed to have 27 different categories to describe the color of the body fluid. Each category was assigned an Arabic numeral and the larger the Arabic numeral, the darker the color of the body fluid. The scoring of sputum coloration was based on the perception of the interviewer who was blinded to the intervention.
Effectiveness as determined by chest X-ray improvement rates | up to 5 days after extubation
  Baseline and follow-up CXRs were taken on the day of extubation and on the 5th day after extubation, respectively, in both groups. Serial changes in CXR were graded as "improved", "no change", or "progressed", as determined by the severity of lung infiltrates, which were defined by two independent chest specialists blinded to the study groupings. If no consistency between two specialists, the grading would be judged by the third chest specialist.

SECONDARY OUTCOMES:
safety as determined by the changes of blood pressures before and after HFCWO | up to 5 days after extubation
  systolic blood pressure (SBP) and diastolic blood pressure (DBP) were recorded before and after each HFCWO treatment by nurses who were unblinded to the study groupings.
safety as determined by the changes of heart rates before and after HFCWO | up to 5 days after extubation
  Heart rates (HR) was recorded before and after each HFCWO treatment by nurses who were unblinded to the study groupings.
safety as determined by the changes of respiratory rates (RR) before and after HFCWO | up to 5 days after extubation
  Respiratory rates (RR) were recorded before and after each HFCWO treatment by nurses who were unblinded to the study groupings.
safety as determined by the changes of oxyhemoglobin saturations by pulse oximetry (SpO2) before and after HFCWO | up to 5 days after extubation
  Oxyhemoglobin saturations by pulse oximetry (SpO2) were recorded before and after each HFCWO treatment by nurses who were unblinded to the study groupings.
tolerance/comfort as determined by Modified Borg Scale (MBS) | up to 5 days after extubation
  MBS was measured before and after treatment in HFCWO group and at the same time in non-HFCWO group by the interviewer who was blinded to the intervention from the day of extubation to the 5th post-extubation day.
tolerance/comfort as determined by Hamilton Anxiety Scale (HAS) | up to 5 days after extubation
  HAS was measured before and after treatment in HFCWO group and at the same time in non-HFCWO group by the interviewer who was blinded to the intervention from the day of extubation to the 5th post-extubation day.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Liang Wu, Ph.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan